CLINICAL TRIAL: NCT03500107
Title: Use of Blue Light Emitting Diode in the Treatment of Women With Bacterial Vaginosis: a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Collaborators: University of Messina (Other); Salvatore Giovanni Vitale M.D. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Centro CAAP
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Vaginosis, Bacterial
Keywords: Blue Light Emitting Diode; Women
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blue LED 401 +/- 5 nm (Experimental): The Blue LED 401 +/- 5 nm will be applied in the participant, in a closed room by a physiotherapist for 1 hour. The apparatus will be supported on a tripod, statically, externally, 5 cm away from the vulva abd vaginal region, with the patient naked, in gynecological stretcher and lithotomy position. The protocol consists of only one session. This part of the study will see if there is bactericidal effect of the blue LED.
  Interventions: Device: Blue Light Emitting Diode (LED) 401 +/- 5nm

INTERVENTIONS:
Device: Blue Light Emitting Diode (LED) 401 +/- 5nm — The participant will be naked, in a gynecological stretcher and lithotomy position, and the apparatus of the LED will be positioned in front of the vulva and vaginal region, 5 cm away, it will be statically, externally, and supported on a tripod. The protocol will consist of only one session.
  Other Names: Questionnaire of anamnesis

SUMMARY:
Bacterial Vaginosis (BV) is a infectious process of the female genitourinary tract, an important health issue due to the high incidence and high rate of recurrence of the infection. Therefore, new therapeutic modalities are sought with the capacity to minimize drug side effects and reduce cases of recurrence of the disease. The objective of this study is to evaluate the clinical and microbiological response of the 401+/- 5nm blue light emitting diode (LED) in the treatment of women with bacterial vaginosis. The group of women with diagnosis of bacterial vaginosis will be submitted to the light therapy. These women will also be submitted to an evaluation and examination by a ginecologist before and after the therapy. There will also be an evaluation of the clinical condition and about the effects of the light through the questionnaire answered before and after participant's treatment. It's expected that the 41 +/- 5nm LED will destroy the VB demonstrated by laboratory examination and also improves the signs and results analyzed by the gynecologist and participants.

DETAILED DESCRIPTION:
A current treatment proposal is the use of blue LED of 401 +/- 5 nm wich is a light that has antimicrobial effect when exposed to endogenous porphyrin of the pathogens. This exposition produces reactive oxygen and it causes cells death with no possibilities of resistance by the bacterium.

ELIGIBILITY:
Inclusion Criteria:

• women with 18 to 65 years old and with diagnosis of bacterial vaginosis

Exclusion Criteria:

• women with injury seen by Pap smear, or in use of pacemaker, with diagnosis or suspicion of neoplasias, with heart diseases, pregnant or with diagnosis of epilepsy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Description of types of cells done by oncology and microflora cytology in women treated by blue LED of 401 +/- 5nm | 15 days
  This exam will be done by the collect of vaginal secretion to analyze types of cells and organisms
Amount of clue cells quantified by fresh cytology in vaginal secretion of women treated by blu LED of 401 +/- 5nm | 10 minutes
  This exam will be done by the collect of vaginal secretion using KOH 10%
Value of vaginal pH measurement in women treated by blue LED | 2 minutes
  This exam will be done by the collect of vaginal secretion using a pH measuring tape to analyse the hydrogen potential in -log 10 [pH+] in women treated by blue LED. It will be used the numeric scale of pH value
Identification of bacterial vaginosis by the culture in vaginal secretion of women treated by blue LED | 15 days
  This exam will be done by the collect of vaginal secretion using a Gram exam / culture for bacteria in women treated by blue LED

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lordelo, Study Director — Centro de Atenção ao Assoalho Pélvico
Locations (1):
- Cebtro de Atebçao ao Assolaho Pévico- Escola Bahiana de Medicina e Saúde Pública, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No